CLINICAL TRIAL: NCT01062594
Title: A Randomised Controlled Trial to Assess the Effect of a Pre-operative Supervised Exercise Programme on Outcome Following Intervention for Abdominal Aortic Aneurysms.
Brief Title: Effect of Pre-operative Exercise in Abdominal Aortic Aneurysms (AAA) Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R0858
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised exercise group (Active Comparator)
  Interventions: Other: Supervised exercise; Other: Role of exercise; Other: Supervised exercise program
- Control group - no exercise (No Intervention)

INTERVENTIONS:
Other: Supervised exercise — Exercise class, this will be performed three times a week with average duration of 40 minutes for 4-6 weeks.
  Arms: Supervised exercise group
Other: Role of exercise — Exercise class, this will be performed three times a week with average duration of 40 minutes for 4-6 weeks.
  Arms: Supervised exercise group
Other: Supervised exercise program — Exercise class, this will be performed three times a week with average duration of 40 minutes for 4-6 weeks.
  Arms: Supervised exercise group

SUMMARY:
An aneurysm is a permanent and localized dilatation of an artery usually more than 50% of its normal diameter. Abdominal Aortic Aneurysms (AAA) is an aneurysm of the main artery of abdomen and affects 5% of men aged 65-74 years. Rupture of an aneurysm is the 10th leading cause of death in white men over 65 years of age in industrial countries. Treatment of asymptomatic AAA is considered when the diameter of an AAA reaches 5.5 cm. There are two treatment options available: conventional open surgical repair or endovascular repair, which is a less invasive mode of treatment. After the operation heart and lung complications are significant in patients undergoing major abdominal surgery. The commonest causes of death are due to heart problems. There are various studies which have shown benefits of pre operative exercise training in patients undergoing orthopaedic, lung and heart bypass surgery. Currently, there is no data available with regards to the effect of pre-operative (before operation) supervised exercise in patients undergoing surgery for an AAA.

The main aim of this study will be to determine whether a pre-operative supervised exercise programme improves post-operative (after operation) outcome, compared to standard treatment.

Patients will be entered in the study once a decision to repair their AAA has been made by the consultant. They will undergo pre-operative assessment and will be divided randomly into two groups. One group will have exercise training for 4-6 weeks before surgery and the other will not. After the operation they will be followed during the post-operative period to determine the presence or absence of complications. It is anticipated that complications will be less in the group which has undertaken exercise training before operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open repair for an asymptomatic peri-renal and infra-renal abdominal aortic aneurysm.
* Patients undergoing Endovascular aneurysm repair (EVAR).
* Able to comply with study protocol.
* Able to give informed consent.

Exclusion Criteria:

* Patients with severe disabling disorders limiting mobility for example severe osteoarthritis.
* Patients undergoing emergency repair of Abdominal Aortic Aneurysm.
* Patients with thoraco abdominal aneurysms.
* Patients unable to communicate in English.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-12; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite outcome including cardiac, respiratory and renal complications | First three months after intervention

SECONDARY OUTCOMES:
Length of ITU/ HDU stay, length of hospital stay (medical/ total), quality of life scores (SF-8 and EURQOL) & death within 30 days of surgery | First three months after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Hull & East Yorkshire Hospitals NHS Trust, Hull, United Kingdom

REFERENCES:
- [Result] Barakat HM, Shahin Y, Khan JA, McCollum PT, Chetter IC. Preoperative Supervised Exercise Improves Outcomes After Elective Abdominal Aortic Aneurysm Repair: A Randomized Controlled Trial. Ann Surg. 2016 Jul;264(1):47-53. doi: 10.1097/SLA.0000000000001609. PMID 26756766
- See also: Publication Link — https://journals.lww.com/annalsofsurgery/fulltext/2016/07000/Preoperative_Supervised_Exercise_Improves_Outcomes.10.aspx